CLINICAL TRIAL: NCT05417152
Title: Evaluation of Repeated, In-Clinic, Self-Imaging by DME Patients Using the Notal Vision Home OCT
Brief Title: Single In-Clinic Encounter With the Notal Vision Home OCT by DME Patients
Status: Completed | Type: Observational
Sponsor: Notal Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C2021.003
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this clinical study the Notal Vision Home OCT (NVHO) Monitoring System will be used to evaluate the ability of patients diagnosed with DME to perform sequential self-images of their eyes with the self-operated NVHO device in a home simulated environment in the doctor's office.

The study population will include up to 30 patients, with DR in at least one eye at the time of enrollment. All subjects will be enrolled at one site in Israel.

DETAILED DESCRIPTION:
Office Visit NOTE: Any planned treatment for DME at the day of the study should be administered after completion of all study-related scans

At the enrollment Office Visit, the exams will be conducted in the following order:

1. Patient will be informed concerning the study and sign the Informed Consent Form (ICF) prior to conduct of any study procedures.
2. Following signing the ICF, subjects will be assigned a Subject ID by a designated staff at the clinical site.
3. The following data will be collected for each study subject:

   1. Date of birth
   2. Gender
   3. Number and type of Anti-VEGF injections and last injection date

3. Refraction correction 4. Snellen BCVA on both eyes on the day of the visit. 5. Eligible eye(s) of the subject will be scanned, non-dilated, with a Zeiss Cirrus OCT device with one (1) acceptable volume scan of each eye being obtained out of up to 3 attempts.

Scanning pattern to be used:

Macular cube, 6X6mm, 128 B-scans per volume scan 6. Eyes of the subject that meet all screening criteria will be enrolled. If both eyes of the subjects meet all screening criteria both eyes will be enrolled.

NOTE: Approximately 90% of the enrolled subjects should have at least one eye with DME at the time of enrollment.

7. The following data will be collected for the study eye(s):

a. Qualifying diagnosis for the study eye from the subject's medical record b. From the subject's medical record, the presence of other ophthalmic conditions including but not limited to: i. Cataract ii. Glaucoma iii. Dry Eye iv. Other macula findings, e.g., epi retinal membrane, macular hole, vitreo-macular traction (VMT)

Following confirmation of subject eligibility, subject will be placed in a room with the NVHO device which has been set up by a technician.

1. The technician will register the subject using the touchscreen of the NVHO device using the subject's CRF number.
2. The subject will perform a self-tutorial. The training flow begins with demonstration clips followed by a practice session. The training flow will be followed by a self-scan that the system uses as a calibration session.
3. Following completion of the training and calibration session, the clinic technician shall set the device for self-scanning flow. The subject will perform four (4) unsupervised self-scans on each study eye with a rest period of ~2 minutes between self-scans.

5. AEs, if applicable, will be collected. 6. Exit subject from the study

ELIGIBILITY:
Inclusion Criteria:

1. Ability to speak, read and understand Hebrew.
2. Ability to understand and agree to contents of informed consent.
3. Eighteen (18) years of age or older at the time of Informed Consent.
4. Subjects diagnosed with DR (Diabetic Retinopathy) in at least one eye, with or without DME
5. Best corrected Visual Acuity of 20/320 (6/96) or better in eyes participating at the study.

Exclusion Criteria:

1. Subjects with dilated pupils.
2. Subjects with other retinal disease requiring steroidal or anti-VEGF injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include up to thirty (30) patients, with DR in at least one eye at the time of enrollment. All subjects will be enrolled at one (1) site in Israel. The subjects must meet all inclusion / exclusion criteria. Approximately 90% of the enrolled subjects should have at least one eye with DME at the time of enrollment.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
NVHO Total Retinal Fluid (TRF) | 5 minutes
  volume (nl) measured by NOA (automatic OCT analyzer)
NVHO Intra-Retinal Fluid (IRF) | 5 minutes
  volume (nl) measured by NOA (automatic OCT analyzer)
NVHO Sub-Retinal Fluid (SRF) | 5 minutes
  volume (nl) measured by NOA (automatic OCT analyzer)
Zeiss Cirrus OCT Total Retinal Fluid (TRF) | 10 minutes
  volume (nl) measured by a human reader
Zeiss Cirrus OCT Intra-Retinal Fluid (IRF) | 10 minutes
  volume (nl) measured by a human reader
Zeiss Cirrus OCT Sub-Retinal Fluid (SRF) | 10 minutes
  volume (nl) measured by a human reader
Scanning session completion status | 5 minutes
  complete/incomplete

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Hashalom, Tel Aviv, Israel